CLINICAL TRIAL: NCT02757963
Title: Implementation of a Screening Tool for Subjects With Benign Prostatic Enlargement/Obstruction to Identify Men >=50 Years Presenting in General Practice With Other Co-morbidities Who Should be Assessed for BPH
Brief Title: Benign Prostatic Hyperplasia (BPH) Screening Tool Case Finding Study in Subjects >=50 Years
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 116114
Record Dates: First submitted 2016-04-28; First posted 2016-05-02 (Estimated); Results first posted 2019-06-24 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Prostatic Hyperplasia
Keywords: Screening tool; International Prostate Symptom Score; Lower urinary tract symptoms; BPO; BPE; Benign prostatic enlargement; Benign prostatic obstruction; LUTS; Benign prostatic hyperplasia; IPSS; BPH
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BPE/BPO screening and IPSS screening tool (Other): Subjects presenting to a GP with a primary complaint other than LUTS will be screened for probable BPH using BPE/BPO screening tool and the IPSS screening tool. Subjects testing positive on the BPE/BPO screening tool or on the IPSS will be enrolled and offered a prostate specific antigen (PSA) test and urinalysis to establish a diagnosis of probable benign prostatic hyperplasia (BPH) (Part I - Visit 1). If the GP determines that the subject has probable BPH (IPSS >=8 and/or BPE/BPO questionnaire >=3 with a PSA >=2 ng per ml), the subject will proceed to Part II and will be scheduled for an urologist assessment and diagnostic tests to confirm or refute a BPH diagnosis and to assess risk of progression of BPH.
  Interventions: Other: Benign prostatic enlargement (BPE)/Benign prostatic obstruction (BPO) screening tool; Other: International Prostate Symptom Score (IPSS) screening tool

INTERVENTIONS:
Other: Benign prostatic enlargement (BPE)/Benign prostatic obstruction (BPO) screening tool — The BPE/BPO screening tool has been developed using the currently recommended Food and Drug Administration (FDA) 2009 guidelines for developing patient-completed questionnaires such as Patient Reported Outcomes. The tool to be used in this study in the General Practice setting has undergone validation in a urology setting to demonstrate the validity of the tool in populations with and without a definite diagnosis of BPH. Subjects who have a positive score on the BPE/BPO screening tool (total score >=3) and meet all other eligibility requirements will be enrolled in Part I of the study.
Other: International Prostate Symptom Score (IPSS) screening tool — The International Prostate Symptom Score (IPSS) score is a validated tool to assess the severity of LUTS symptoms, and has similarly been used for assessing symptomatic efficacy of treatments for BPH. Subjects who have a positive score on the IPSS tool (score >=8) and meet all other eligibility requirements will be enrolled in Part I of the study.

SUMMARY:
This non-randomized, interventional study will be conducted in a general practice setting to assess the utility of a benign prostatic enlargement (BPE)/benign prostatic obstruction (BPO) screening tool in conjunction with prostate specific antigen (PSA) in finding men confirmed to have BPH on full urologist assessment of diagnostic test results. The tool may help a General Practitioners (GP) to identify subjects who may have BPH for further tests and improve the speed of referrals to specialists when this is appropriate. The utility of the screening tool will be compared to the validated tool in wide clinical use, the International Prostate Symptom Score (IPSS). This study does not have any formal hypothesis in terms of the primary and secondary endpoint proportions. A BPE/BPO screening tool identifies lower urinary tract symptoms (LUTS) probably due to BPH in men not yet presenting with LUTS. The results of this screening tool will be used for further investigation. All subjects testing positive on the BPE/BPO screening tool (score >=3) tool or on the IPSS (score >=8) will be enrolled and offered a PSA test and urinalysis to establish a diagnosis of probable BPH (Part I-Visit 1). The GP may perform a digital rectal examination (DRE) which will be repeated by the urologist to confirm the diagnosis and to rule out an abnormality suggesting prostate cancer. The GP will make a diagnosis of probable BPH based upon screening results and lab tests which suggest that they are related to BPH and not other causes of such symptoms. The GP will phone the subject to report yes or no for probable BPH Part II (Visit 2). If the subject has probable BPH, the GP will schedule the subject for Visit 3 with an urologist. If the subject does not have probable BPH, then it will be considered that the subject has completed the study. Subjects that proceed to Part II (Visit 3) will be scheduled for a urology assessment performed by an urologist. This assessment includes a DRE and a brief physical exam and review of the PSA test, for a confirmatory diagnosis of BPH and estimation of risk of progression of BPH. Approximately 1,500 subjects presenting to a GP for reasons unrelated to this study will be screened for probable BPH to yield 500 subjects being referred to an urologist. The duration of the study will be 1 week (+/- 4 days) and up to 6 weeks to allow for GP and urologist visit scheduling.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to (>=) 50 years of age at the time of signing the informed consent form.
* Male.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and protocol.
* Present in a General Practice setting for a reason unrelated to this study.
* Positive IPSS score >=8 and/or positive BPE/BPO screening tool score >=3.

Exclusion Criteria:

* History of BPH for which they have received test procedures, medical intervention and/or medicine.
* History of prostate-related LUTS for which they have received test procedures, medical intervention and/or medicine.
* History of prostatic surgery (including transurethral resection of the prostate (TURP), balloon dilatation, thermotherapy, and/or stent replacement) or other invasive or minimally invasive procedures to treat BPH.
* Has other conditions that may cause urinary symptoms (e.g., neurogenic bladder, bladder neck contracture, urethral stricture, bladder malignancy, acute or chronic prostatitis, or acute or chronic urinary tract infections, etc.).
* History or evidence of prostate cancer (e.g., positive biopsy or ultrasound, suspicious DRE and/or rising PSA).
* Current or prior use of the following: 5alpha-reductase inhibitors (finasteride or dutasteride); anti-cholinergics (e.g. oxybutynin, propantheline, tolterodine, solifenacin, darifenacin, mirabegron) alpha-adrenoreceptor blockers (i.e., indoramin, prazosin, terazosin, tamsulosin, alfuzosin, doxazosin and silodosin), herbal products for urinary symptoms; Use of any investigational study drug within 30 days or 5 half-lives of the drug in question, (whichever is longer), preceding the first study visit.
* Use within previous 30 days at Visit 1 of: phosphodiesterase type 5 inhibitor (PDE-5) inhibitors for erectile dysfunction; anabolic steroids

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1679 (Actual)
Dates: Start 2016-05-12 (Actual); Primary Completion 2017-02-27 (Actual); Study Completion 2017-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (42):
- France (8):
  - GSK Investigational Site, Aigrefeuille-sur-Maine
  - GSK Investigational Site, Grenay
  - GSK Investigational Site, Haute-Goulaine
  - GSK Investigational Site, La Montagne
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Rosiers-d'Égletons
  - GSK Investigational Site, Rouen
  - GSK Investigational Site, Thouars
- Germany (9):
  - GSK Investigational Site, Weinheim, Baden-Wurttemberg
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Flörsheim, Hesse
  - GSK Investigational Site, Buchholz, Lower Saxony
  - GSK Investigational Site, Dippoldiswalde, Saxony
  - GSK Investigational Site, Freital, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Magdeburg
- Italy (6):
  - GSK Investigational Site, Aradeo, Apulia
  - GSK Investigational Site, Cutrofiano (LE), Apulia
  - GSK Investigational Site, Galatina (LE), Apulia
  - GSK Investigational Site, Ruffano (LE), Apulia
  - GSK Investigational Site, Civitella Paganico (GR), Tuscany
  - GSK Investigational Site, Grosseto, Tuscany
- Russia (14):
  - GSK Investigational Site, Arkhangelsk
  - GSK Investigational Site, Ivanovo
  - GSK Investigational Site, Izhevsk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Naro-Fominsk
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, Odintsovo
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Saint Petesburg
  - GSK Investigational Site, Smolensk
  - GSK Investigational Site, St'Petersburg
  - GSK Investigational Site, Tomsk
  - GSK Investigational Site, Ulyanovsk
  - GSK Investigational Site, Yaroslavl
- Spain (5):
  - GSK Investigational Site, Bormujo (Sevilla)
  - GSK Investigational Site, Cadiz
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study is available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (copy the URL below to your browser)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://www.clinicalstudydatarequest.com/Posting.aspx?ID=20742

REFERENCES:
- [Background] Tubaro A, Niero M, Adalig B, Lulic Z, Plastino J, Kimbrough C, Manyak MJ. Evaluation of a 3-item screening tool to identify men with benign prostatic enlargement/obstruction in a primary care cohort. Minerva Urol Nephrol. 2022 Feb;74(1):85-92. doi: 10.23736/S2724-6051.20.03834-5. Epub 2020 Sep 29. PMID 32993275

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1658 male participants, >=50 years of age, with reasons not related to lower urinary tract symptoms (LUTS) were included in evaluable Population. The study was conducted at 47 centers in 5 countries; 8 centers in France, 9 centers in Germany, 6 centers in Italy, 18 centers in Russia and 6 centers in Spain.
Pre-assignment Details: A total of 2343 male participants were screened for probable Benign prostatic hyperplasia (BPH). Of these, 1679 participants were enrolled, 1658 participants were included in the evaluable population. 21 participants progressed in the study but were found to have not met eligibility criteria. Overall, 561 participants completed all 3 visits.
Groups:
- IPSS >=8 or BPE/BPO >=3: Participants were screened using the Benign prostatic enlargement (BPE)/ benign prostatic obstruction (BPO) and International Prostate Symptom Score (IPSS) screening tools. Participants with positive responses (i.e. met entry criteria, including positive IPSS score >= 8 and/or BPE/BPO score >= 3) were enrolled and proceeded to Part I (GP Assessment). Participants with probable BPH [PSA>= 2 Nano gram per milliliter (ng/mL)] proceeded to Part II and were scheduled for a urologist assessment which was to confirm or refute a diagnosis of BPH and to estimate whether the participant is at risk of progression of BPH.
Period: Overall Study
Arm/Group | IPSS >=8 or BPE/BPO >=3
Started | 1658
Completed | 561
Not Completed | 1097
Not completed — Adverse Event | 3
Not completed — Reached Stopping Criteria | 1054
Not completed — Lost to Follow-up | 5
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 34

BASELINE CHARACTERISTICS:
Groups:
- IPSS >=8 or BPE/BPO >=3: Participants were screened using the BPE/BPO and IPSS screening tools. Participants with positive responses (i.e. met entry criteria, including positive IPSS score >=8 and/or BPE/BPO score >=3) were enrolled and proceeded to Part I (GP Assessment). Participants with probable BPH (PSA>=2 ng/mL) proceeded to Part II and were scheduled for a urologist assessment which was to confirm or refute a diagnosis of BPH and to estimate whether the participant is at risk of progression of BPH.
Arm/Group | IPSS >=8 or BPE/BPO >=3
Number analyzed (Participants) | 1658
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.8 (8.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1658
Race/Ethnicity, Customized [Number; unit: Participants] — Population: Race information was not collected for 99 participants who were enrolled in the study in France.
  Participants
    African American/African Heritage: number analyzed (Participants) | 1559
    African American/African Heritage | 2
    Asian - Central/South Asian Heritage: number analyzed (Participants) | 1559
    Asian - Central/South Asian Heritage | 2
    White - Arabic/ North African Heritage: number analyzed (Participants) | 1559
    White - Arabic/ North African Heritage | 2
    White - White/ Caucasian/European Heritage: number analyzed (Participants) | 1559
    White - White/ Caucasian/European Heritage | 1550
    White - Mixed Race: number analyzed (Participants) | 1559
    White - Mixed Race | 1
    Mixed Race: number analyzed (Participants) | 1559
    Mixed Race | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Men With Confirmed Diagnosis of BPH
Description: Confirmed diagnosis of BPH was based on full urologist diagnostic testing with a positive result on the BPE/BPO screening tool (score >=3) and serum PSA >=2 ng/mL. The BPE/BPO questionnaire consists of three questions each with a score ranging from 0= never experienced to 5= almost always experienced. Participants with probable BPH underwent full urologist diagnostic testing, which included review of medical history, symptoms and previous tests, brief physical examination, Digital rectal examination (DRE). Proportion of participants was calculated by dividing number of participants with a positive result on the BPE/BPO screening tool (Score >= 3) and a diagnosis of BPH by the urologist (Numerator) by number of participants with a positive result on the BPE/BPO screening tool (Score >= 3) and a BPH assessment by the urologist (Denominator). 95% confidence interval on the proportion was calculated by using the exact (Clopper-Pearson) method.
Time Frame: Up to 6 weeks
Population: All Evaluable Subject Population comprised of all participants who meet the entry criteria, including a positive IPSS screening result (score >=8) and/or a positive BPE/BPO screening result (score >=3).
Measure: Count of Participants; unit: Participants
Groups:
- BPE/BPO >=3: Participants were screened using the BPE/ BPO screening tools. Participants with a positive response to this tool (i.e. Participants met entry criteria, including a positive BPE/BPO score >= 3) were enrolled and proceeded to Part I (GP Assessment) of the study. Participants with probable BPH (PSA>= 2 ng/mL) proceeded to Part II and were scheduled for the urologist assessment to confirm diagnosis of BPH and to estimate whether the participant was at risk of progression of BPH
Arm/Group | BPE/BPO >=3
Number analyzed (Participants) | 1249
Participants
  Numerator | 386
  Denominator | 437
Statistical Analysis 1: Comparison: BPE/BPO >=3; Test type: Other; Proportion = 0.883, 95% CI 2-sided [0.849 to 0.912] — Proportion = Numerator / Denominator. 95% confidence interval on the proportion is calculated by using the exact (Clopper-Pearson) method

2. Secondary Outcome: Number of Men That Are Confirmed to Have BPH Based on Full Urologist Assessment of Diagnostic Test Results Among Men With a Positive Result on the IPSS, BPE/BPO and IPSS, and BPE/BPO or IPSS Screening Tools and Serum PSA >=2 ng/mL
Description: Confirmed diagnosis of BPH was based on full urologist diagnostic testing with a positive result on the IPSS, BPE/BPO and IPSS, BPE/BPO or IPSS screening tools and serum PSA >=2 ng/mL. The BPE/BPO questionnaire consists of three questions each with a score ranging from 0= never experienced to 5= almost always experienced. IPSS tool is used to assess the severity of LUTS symptoms with a score ranging from 0= never experienced to 5= almost always experienced. Participants with probable BPH underwent full urologist diagnostic testing, which included review of medical history, symptoms and previous tests, brief physical examination, DRE. Proportion of participants was calculated by dividing number of participants with a positive result on the screening tool and a diagnosis of BPH by the urologist (Numerator) by number of participants with a positive result on the screening tool and a BPH assessment by the urologist(Denominator).
Time Frame: Up to 6 weeks
Population: All Evaluable Subjects Population
Measure: Count of Participants; unit: Participants
Groups:
- IPSS >=8: Participants were screened using the IPSS screening tool. Participants with a positive response to this tool (i.e. Participants met entry criteria, including a positive IPSS score >=8) were enrolled and proceeded to Part I (GP Assessment) of the study. Participants with probable BPH (PSA >=2 ng/mL) proceeded to Part II and were scheduled for the urologist assessment to confirm diagnosis of BPH and to estimate whether the participant was at risk of progression of BPH.
- IPSS >=8 and BPE/BPO >=3: Participants were screened using the BPE/BPO and IPSS screening tools. Participants with positive responses to these tools (i.e. Participants met entry criteria, including a positive IPSS score >=8 and BPE/BPO score >=3) were enrolled and proceeded to Part I (GP Assessment) of the study. Participants with probable BPH (PSA >=2 ng/mL) proceeded to Part II and were scheduled for the urologist assessment to confirm diagnosis of BPH and to estimate whether the participant was at risk of progression of BPH
- IPSS >=8 or BPE/BPO >=3: Participants were screened using the BPE/BPO and IPSS screening tools. Participants with positive responses to these tools (i.e. Participants met entry criteria, including a positive IPSS score >=8 or BPE/BPO score >=3) were enrolled and proceeded to Part I (GP Assessment) of the study. Participants with probable BPH (PSA >=2 ng/mL) proceeded to Part II and were scheduled for the urologist assessment to confirm diagnosis of BPH and to estimate whether the participant was at risk of progression of BPH
Arm/Group | IPSS >=8 | IPSS >=8 and BPE/BPO >=3 | IPSS >=8 or BPE/BPO >=3
Number analyzed (Participants) | 1558 | 1149 | 1658
Participants
  Numerator | 471 | 367 | 490
  Denominator | 537 | 413 | 561
Statistical Analysis 1: Comparison: IPSS >=8; For Arm IPSS >=8; Test type: Other; Proportion = 0.877, 95% CI 2-sided [0.846 to 0.904] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: IPSS >=8 and BPE/BPO >=3; For Arm IPSS >=8 and BPE/BPO >=3; Test type: Other; Proportion = 0.889, 95% CI 2-sided [0.854 to 0.917] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: IPSS >=8 or BPE/BPO >=3; For Arm IPSS >=8 or BPE/BPO >=3; Test type: Other; Proportion = 0.873, 95% CI 2-sided [0.843 to 0.900] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Number of Men That Are Confirmed to be at Risk for BPH Progression Based Upon Full Urologist Assessment Among Men With a Positive Result on the BPE/BPO, IPSS, BPE/BPO and IPSS, and BPE/BPO or IPSS Screening Tools and Serum PSA >=2 ng/mL
Description: Confirmed risk for BPH was based on full urologist diagnostic testing with a positive result on the BPE/BPO and/or IPSS screening tool and probable GP BPH diagnosis. The BPE/BPO questionnaire consists of 3 questions each with a score from 0= never experienced to 5= almost always experienced. IPSS tool is used to assess the severity of LUTS symptoms with a score from 0= never experienced to 5= almost always experienced. Participants with probable BPH underwent full urologist diagnostic testing, which included review of medical history, symptoms and previous tests, physical examination, DRE. Participants with PSA >=2.0 ng/mL and other tests were considered as at risk for BPH. Proportion of participants was calculated by dividing number of participants with a positive result on the screening tool and diagnosis of BPH progression risk (Numerator) by number of participants with a positive result on the screening tool and a BPH progression risk assessment by the urologist (Denominator).
Time Frame: Up to 6 weeks
Population: All Evaluable Subjects Population
Measure: Count of Participants; unit: Participants
Groups:
- IPSS >=8: Participants were screened using the IPSS screening tool. Participants with a positive response to this tool (i.e. Participants met entry criteria, including a positive IPSS score >= 8) were enrolled and proceeded to Part I (GP Assessment) of the study. Participants with probable BPH (PSA >= 2 ng/mL) proceeded to Part II and were scheduled for the urologist assessment to confirm diagnosis of BPH and to estimate whether the participant was at risk of progression of BPH.
- BPE/BPO >=3: Participants were screened using BPE/BPO screening tool. Participants with a positive response to this tool (i.e. Participants met entry criteria, including a positive BPE/BPO score >=3) were enrolled and proceeded to Part I (GP Assessment) of the study. Participants with probable BPH (PSA >=2 ng/mL) proceeded to Part II and were scheduled for the urologist assessment to confirm diagnosis of BPH and to estimate risk of progression of BPH
- IPSS >=8 and BPE/BPO >=3: Participants were screened using the BPE/BPO and IPSS screening tools. Participants with positive responses to these tools (i.e. Participants met entry criteria, including a positive IPSS score >= 8 and BPE/BPO score >= 3) were enrolled and proceeded to Part I (GP Assessment) of the study. Participants with probable BPH (PSA >= 2 ng/mL) proceeded to Part II and were scheduled for the urologist assessment to confirm diagnosis of BPH and to estimate whether the participant was at risk of progression of BPH
- IPSS >=8 or BPE/BPO >=3: Participants were screened using the BPE/BPO and IPSS screening tools. Participants with positive responses to these tools (i.e. Participants met entry criteria, including a positive IPSS score >= 8 or BPE/BPO score >= 3) were enrolled and proceeded to Part I (GP Assessment) of the study. Participants with probable BPH (PSA >= 2 ng/mL) proceeded to Part II and were scheduled for the urologist assessment to confirm diagnosis of BPH and to estimate whether the participant was at risk of progression of BPH
Arm/Group | IPSS >=8 | BPE/BPO >=3 | IPSS >=8 and BPE/BPO >=3 | IPSS >=8 or BPE/BPO >=3
Number analyzed (Participants) | 1558 | 1249 | 1149 | 1658
Participants
  Numerator | 424 | 350 | 333 | 441
  Denominator | 471 | 386 | 367 | 490
Statistical Analysis 1: Comparison: IPSS >=8; For Arm IPSS >=8; Test type: Other; Proportion = 0.900, 95% CI 2-sided [0.870 to 0.926] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: BPE/BPO >=3; For Arm BPE/BPO >=3; Test type: Other; Proportion = 0.907, 95% CI 2-sided [0.873 to 0.934] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: IPSS >=8 and BPE/BPO >=3; For Arm IPSS >=8 and BPE/BPO >=3; Test type: Other; Proportion = 0.907, 95% CI 2-sided [0.873 to 0.935] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: IPSS >=8 or BPE/BPO >=3; For Arm PSS >=8 or BPE/BPO >=3; Test type: Other; Proportion = 0.900, 95% CI 2-sided [0.870 to 0.925] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Number of Men That Are Diagnosed With Probable BPH as Assessed by the GP Among Men With a Positive Result on the BPE/BPO, IPSS, BPE/BPO and IPSS, and BPE/BPO or IPSS Screening Tools
Description: Diagnosis of probable BPH was based on GP assessment among men with a positive result on the BPE/BPO and/or IPSS screening tool. The BPE/BPO questionnaire consists of 3 questions each with a score from 0= never experienced to 5= almost always experienced. IPSS tool is used to assess the severity of LUTS symptoms with a score from 0= never experienced to 5= almost always experienced. Probable BPH is the presumptive diagnosis of urinary tract obstruction from an enlarged prostate based on clinical symptoms and findings where urinary symptoms are not apparently related to any other cause. Participants underwent GP assessment and lab result review by GP. Participants with PSA >=2 ng/mL were assessed for probable BPH. Proportion of participants was calculated by dividing number of participants with a positive result on the screening tool and diagnosis of probable BPH (Numerator) by number of participants with a positive result on the screening tool and a BPH assessment by GP (Denominator).
Time Frame: Up to 6 weeks
Population: All Evaluable Subjects Population
Measure: Count of Participants; unit: Participants
Groups:
- BPE/BPO >=3: Participants were screened using BPE/BPO screening tools. Participants with a positive response to this tool (i.e. Participants met entry criteria, including a positive BPE/BPO score >=3) were enrolled and proceeded to Part I (GP Assessment) of the study. Participants with probable BPH (PSA >=2 ng/mL) proceeded to Part II and were scheduled for the urologist assessment to confirm diagnosis of BPH and to estimate risk of progression of BPH
- IPSS >= 8 or BPE/BPO >=3: Participants were screened using the BPE/BPO and IPSS screening tools. Participants with positive responses to these tools (i.e. Participants met entry criteria, including a positive IPSS score >=8 or BPE/BPO score >=3) were enrolled and proceeded to Part I (GP Assessment) of the study. Participants with probable BPH (PSA >=2 ng/mL) proceeded to Part II and were scheduled for the urologist assessment to confirm diagnosis of BPH and to estimate whether the participant was at risk of progression of BPH
Arm/Group | IPSS >=8 | BPE/BPO >=3 | IPSS >=8 and BPE/BPO >=3 | IPSS >= 8 or BPE/BPO >=3
Number analyzed (Participants) | 1558 | 1249 | 1149 | 1658
Participants
  Numerator | 556 | 453 | 428 | 581
  Denominator | 1538 | 1232 | 1135 | 1635
Statistical Analysis 1: Comparison: IPSS >=8; For Arm IPSS >=8; Test type: Other; Proportion = 0.362, 95% CI 2-sided [0.337 to 0.386] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: BPE/BPO >=3; For Arm BPE/BPO >=3; Test type: Other; Proportion = 0.368, 95% CI 2-sided [0.341 to 0.395] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: IPSS >=8 and BPE/BPO >=3; For Arm IPSS >=8 and BPE/BPO >=3; Test type: Other; Proportion = 0.377, 95% CI 2-sided [0.349 to 0.406] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: IPSS >= 8 or BPE/BPO >=3; For Arm IPSS >=8 or BPE/BPO >=3; Test type: Other; Proportion = 0.355, 95% CI 2-sided [0.332 to 0.379] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Summary of Agreement Between BPE/BPO and IPSS Screening Tools
Description: Agreement between the IPSS and BPE/BPO tools had to utilize the screened population, as the evaluable population did not include any participants with IPSS <8 and BPE/BPO<3. All screened participants with IPSS and BPE/BPO results were utilized (2327 of the 2343 participants had IPSS and BPE/PO results). There were 16 participants (2343 minus 2327) in the screened population without IPSS and BPE/BPO results, and hence were not included in the calculation of the Kappa statistic. Kappa statistic values of <0 were characterized as no agreement, 0 to 0.20 as slight, 0.21 to 0.40 as fair, 0.41 to 0.60 as moderate, 0.61 to 0.80 as substantial, and 0.81 to 1.00 as almost perfect agreement. The 95% confidence interval for the Kappa statistic is based on the asymptotic standard error.
Time Frame: Day 1
Population: All Screened Subjects Population comprised of all participants who were screened for eligibility. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Count of Participants; unit: Participants
Groups:
- All Screened Subjects: All the participants who signed informed consent form and were screened for eligibility were included in this arm
Arm/Group | All Screened Subjects
Number analyzed (Participants) | 2327
Participants | 1812
Statistical Analysis 1: Comparison: All Screened Subjects; Test type: Other; Kappa statistic = 0.55, 95% CI 2-sided [0.51 to 0.58]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and serious adverse events (SAEs) were collected from screening (Visit 1) through 6 weeks
Description: On-therapy SAEs and non-serious AEs are reported for members of All Evaluable Subjects Population which comprised of all participants who met the entry criteria, including a positive IPSS screening result (score >=8) and/or a positive BPE/BPO screening result (score >=3)
Groups:
- IPSS >= 8 or BPE/BPO >= 3: Participants were screened using the BPE/BPO and IPSS screening tools. Participants with positive responses to these tools (i.e. Participants met entry criteria, including a positive IPSS score >= 8 or BPE/BPO score >= 3) were enrolled and proceeded to Part I (GP Assessment) of the study. Participants with probable BPH (PSA >= 2 ng/mL) proceeded to Part II and were scheduled for the urologist assessment to confirm diagnosis of BPH and to estimate whether the participant was at risk of progression of BPH
Arm/Group | IPSS >= 8 or BPE/BPO >= 3
All-Cause Mortality (participants affected / at risk) | 1/1658
Serious Adverse Events (participants affected / at risk) | 9/1658
Other Adverse Events (participants affected / at risk) | 0/1658
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IPSS >= 8 or BPE/BPO >= 3 (N=1658)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
Atrial flutter (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Sudden death (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-01-18): https://cdn.clinicaltrials.gov/large-docs/63/NCT02757963/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-20): https://cdn.clinicaltrials.gov/large-docs/63/NCT02757963/SAP_001.pdf